CLINICAL TRIAL: NCT02772796
Title: An Open-label, Single-dose, Pharmacokinetic Study of SENS-218 in Healthy Adult, Caucasian Subjects.
Brief Title: A Single Dose PK Study of SENS-218 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simbec Research (Industry)
Collaborators: Sensorion SA (Unknown)
Responsible Party: Principal Investigator, Girish Sharma, MBBS, Simbec Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RD 716/33020
Record Dates: First submitted 2016-04-25; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Inner Ear Diseases
Keywords: Pharmacokinetics; Healthy Volunteer Study
MeSH Terms: conditions — Labyrinth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENS-218 (Experimental): 2 x 10 mg administered once on Day 1.
  Interventions: Drug: SENS-218

INTERVENTIONS:
Drug: SENS-218 — Oral Administration

SUMMARY:
This study is to aid the development for the use of SENS-218 outside its marketed therapeutic indications. SENS-218 is available in Asia and is marketed as an anti-emetic (Anti-sickness) drug often prescribed after exposure to chemotherapy. Chemotherapy exposure can often induce nausea and/or vomiting.

The study only involves the one drug, referred to as SENS-218 in this study. The purpose of the study is to support the development of use of SENS-218 in non-Asian population.

The key objective of this study is to identify the pharmacokinetic (PK) parameters of the drug in healthy Caucasian population. The PK refers to what the body does to the body, for example, how quickly the drug is absorbed into the blood stream.

The population who are eligible to take part in the study are healthy male and female, non-smoking volunteers, aged between 18 and 50 years, as determined by screening tests at Simbec.

Participation in the trial will last for about 3 weeks (from first screening visit to final end of study visit).

DETAILED DESCRIPTION:
This study consists of a screening visit, 1 treatment period and a post study visit.

These are outlined below:

Screening visit ( Day -14 to Day -1)

- Ensure subjects are eligible for the study.

Treatment period 1 -If all screening assessments are satisfactory, subjects will be invited to attend Simbec to take part in the study. The treatment period consists of 2 overnight stays (Day -1 until the morning of Day 2). One return visit is required at the 48 hour point post dose on Day 3.

Post study visit

-Subjects will be asked to attend Simbec 5-7 days after administration of the last dose for a post study visit. If you are withdrawn from the study, you will still be asked to attend for an end of study assessment.

Subjects may be asked to return again if we need to follow you up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian males and females (non-pregnant/non-lactating) between 18 and 50 years of age.
2. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use 2 effective methods of contraception, from first dose until 3 months afterwards (i.e., until 3 months after taking IMP).
3. Female subject of non-child bearing potential with with negative pregnancy test at the screening visit.

   For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy) and levels of follicle stimulating hormone (FSH) falling within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the Investigator following consultation with the Sponsor's Responsible Physician.
4. Male subject willing to use 2 effective methods of contraception, (unless anatomically sterile) from first dose until 3 months afterwards (i.e., until 3 months after taking IMP).
5. Subject with a body mass index (BMI) of 18-30 kg/m2. BMI = body weight (kg)/height (m)2.
6. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days of the first dose.
7. Subject with a negative urinary drugs of abuse screen, determined within 14 days of the first dose (a positive alcohol result may be repeated at the discretion of the Investigator).
8. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
9. Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 14 days of the first dose.
10. Subject with no clinically significant abnormalities in blood pressure or pulse determined within 14 days of the first dose.
11. Subject is a non-smoker or ex-smoker who has not smoked in the last 3 months (determined by urine cotinine < 500 ng/mL at screening visit).
12. Subject is available to complete the study (including all follow-up visits) and comply with study restrictions.
13. Subject satisfies a medical examiner about their fitness to participate in the study.
14. Subject provides written informed consent to participate in the study.

Exclusion Criteria:

1. Subject with a clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Subject in receipt of regular medication (with the exception of contraception) within 14 days of the first dose that may have an impact on the safety and objectives of the study (Investigator's discretion).
3. Subject with evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. Subjects with any renal (serum creatinine (CREAT) level > 1.5 fold above the upper limit of normal (ULN)) or liver insufficiency (alkaline phosphatase (ALP) level > 1.2 fold above ULN, gamma glutamyl transferase (GGT), aspartate transaminase (AST), or alanine transaminase (ALT) level > 2.5 fold above ULN, and total bilirubin (BIL-T) level > 1.5 fold above ULN).
5. Subject with history of, or family history (immediate relative) of, long QT syndrome or Torsade de Pointes or symptomatic bradycardia.
6. Subject with clinically significant history of previous allergy / sensitivity to SENS-218 or its excipients or other 5-hydroxytryptophan3 (5-HT3) receptor antagonists.
7. Subject with a clinically significant history of drug or alcohol abuse.
8. Subject with inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
9. Subject participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
10. Subject donated 450 mL or more blood within the previous 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cmax - Max plasma concentration of SENS-218 in healthy adults | 0 to 48 hours.
Tmax -Time taken to reach Cmax for SENS-218 in healthy adults | 0 to 48 hours.
kel - elimination rate constant of SENS-218 in healthy adults | 0 to 48 hours.
t1/2 - Terminal Elimination half life of SENS-218 in healthy adults | 0 to 48 hours
AUC0-t - area under the concentration-time curve (AUC) from the time of dosing to last measurable concentration of SENS-218 in healthy adults. | 0 to 48 hours
AUC0-inf - the AUC extrapolated to infinity of SENS-218 in healthy | 0 to 48 hours
CL/F - clearance, calculated as dose/AUC0-inf of SENS-218 in healthy adults. | 0 to 48 hours
MRT - Mean residence time of SENS-218 in healthy adults | 0 to 48 hours

SECONDARY OUTCOMES:
12-lead ECGs | Day 1 until post study (5 to 7 days following IMP administration)
  12-lead ECG assessments: Heart rate, PR interval, QRS width, QT interval and QT interval corrected using Bazett's formula (QTcB).
Vitals signs | Day 1 until post study (5 to 7 days following IMP administration)
  Vital signs assessments: Systolic/diastolic blood pressure and pulse rate and oral body temperature. corrected using Bazett's formula (QTcB).
Physical examination | Day 1 until post study (5 to 7 days following IMP administration)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MBBS, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: Undecided